CLINICAL TRIAL: NCT01743599
Title: Retrograde Ejaculation and Sexual Dysfunction in Men With Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Jens Fedder, Professor, Consultant, Ph.D., Odense University Hospital
Other Study IDs: Lab.Reprod.Biol.-Horsens-01
Record Dates: First submitted 2012-11-27; First posted 2012-12-06 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Diabetic men
- Non-diabetic men

SUMMARY:
Diabetic men and controls are examined for retrograde ejaculation, and erectile dysfunction is registered with a validated questionaire (International Index of Erectile Function-15). Concentration, total number of sperm and motility is determined in freshly delivered ejaculates and postejaculatory urine. Our hypothetis is that diabetics exhibit significantly higher rate of retrograde ejaculation than healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Men 30-55 years of age
* Men registered in a Diabetic Biobank including 6000 diabetics and 6000 controls

Exclusion Criteria:

* Men who do not understand Danish

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Diabetic men and non-diabetic men in Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2008-02; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Retrograde ejaculation (a minimum of a total of 1 million sperm in postejaculatory urine) | The examination program for each patient was finished within one day.

SECONDARY OUTCOMES:
Erectile dysfunction | The examination program (including a questionaire on erectile dysfunction) for each patient was finished within one day.

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Clinic, Odense University Hospital, Odense, Denmark

REFERENCES:
- [Result] Fedder J, Kaspersen MD, Brandslund I, Hojgaard A. Retrograde ejaculation and sexual dysfunction in men with diabetes mellitus: a prospective, controlled study. Andrology. 2013 Jul;1(4):602-6. doi: 10.1111/j.2047-2927.2013.00083.x. Epub 2013 Apr 18. PMID 23606485